CLINICAL TRIAL: NCT01567306
Title: Phase II, Multicenter, Randomized, Double Blind Study, With Subcutaneous Immunotherapy At Different Doses, in Parallel Groups and Placebo-Controlled, in Patients With Rhinoconjunctivitis ± Asthma Sensitized to Phleum Pratense
Brief Title: Phase II Trial With Subcutaneous Immunotherapy in Patients Sensitized to Phleum Pratense
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-PHL-P2-001; 2011-000814-21 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergy; Allergic rhinoconjunctivitis; Subcutaneous Immunotherapy; Phleum pratense pollen extract
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Allergovac Depot Group 1 Active (Experimental)
  Interventions: Biological: Allergovac Depot
- Allergovac Depot Group 2 Active (Experimental)
  Interventions: Biological: Allergovac Depot
- Allergovac Depot Group 3 Active (Experimental)
  Interventions: Biological: Allergovac Depot
- Allergovac Depot Group 4 Active (Experimental)
  Interventions: Biological: Allergovac Depot
- Allergovac Depot Group 5 Active (Experimental)
  Interventions: Biological: Allergovac Depot
- Placebo - Group 6 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allergovac Depot — Increasing dosages till the maintenance dose of 0.25 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Allergovac Depot Group 1 Active
Biological: Allergovac Depot — Increasing dosages till the maintenance dose of 0.5 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Allergovac Depot Group 2 Active
Biological: Allergovac Depot — Increasing dosages till the maintenance dose of 1SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Allergovac Depot Group 3 Active
Biological: Allergovac Depot — Increasing dosages till the maintenance dose of 2 SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Allergovac Depot Group 4 Active
Biological: Allergovac Depot — Increasing dosages till the maintenance dose of 4SPT is reached. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Allergovac Depot Group 5 Active
Biological: Placebo — Increasing volumes of placebo. Afterwards, 3 maintenance doses are given at 4-weekly intervals.
  Other Names: Allergovac
  Arms: Placebo - Group 6

SUMMARY:
Based on EMA (European Medicines Agency) new guidelines on the clinical development of products for immunotherapy for the treatment of allergic diseases the aim of this study is to establish a dose-response relationship for clinical efficacy of Phleum pratense pollen extract subcutaneous vaccine.

DETAILED DESCRIPTION:
In adherence to EMA guidelines, the Phase I Clinical trial was carried out using Phleum pratense extract in depot presentation using 3 different dose escalation scheme. The objective was to compare tolerance and safety of the three dose escalation scheme as well as to determine the maximum dose tolerated by the population.

Once the range of tolerated doses was established, and following the strict norms of the EMA, a Phase II dose response clinical trial was designed wherein the efficacy of subcutaneous immunotherapy in depot presentation could be compared in 5 different doses. One of these doses will be the MTD established by the population in the first study, another will be lower than this dose, and three will be greater than it. The dose escalation scheme to be tested was chosen based on the results of the aforementioned clinical trial. As dictated by EMA norms, a control placebo will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the Informed Consent Form.
2. Patients must be between 18 and 60 years of age.
3. Patients with seasonal allergic rhinoconjunctivitis produced by Phleum pratense during at least 2 years prior to participating in the study. Although the pathology being studied is allergic rhinoconjunctivitis, patients who have concomitant mild or moderate asthma may be included.
4. Patients who have had a skin prick test result equal or more than 3 mm in diameter against Phleum pratense.
5. Patients who have specific IgE equal or more than class 2 (CAP/PHADIA) to Phleum pratense.
6. Patients will preferably be monosensitized to Phleum pratense. Polysensitized patients may only be included in the study if their other sensitizations are produced by:

   * Overlapping seasonal pollens which are cross-reactive with Phleum pratense.
   * Pollens whose seasons do not overlap with Phleum pratense and which are not expected to produce symptoms during the study period.
   * Other allergens which are not expected to produce symptoms during the study period.
7. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.
8. Furthermore, women of child-bearing potential must agree to use adequate contraceptive methods during this study if they are sexually active.

Exclusion Criteria:

1. Patients with stable and continued use of allergy medication during the 2 weeks prior to their inclusion in the study.
2. Patients sensitized to allergens with overlapping seasons but which are not cross-reactive with Phleum pratense and with specific IgE levels equal or less than class 2 CAP/PHADIA.
3. Patients who have received immunotherapy in the 5 years prior to the study against either the allergen being tested or an allergen which is cross-reactive, or who are currently receiving immunotherapy for any other allergen.
4. Patients with severe asthma or FEV1 < 70% or with asthma which requires treatment with inhaled or systemic corticoids at the time of the study or in the 8 weeks immediately prior to the onset of treatment.
5. Patients with immunological, cardiac, renal or hepatic diseases or any with any other illness which the investigators deem may interfere with the study.
6. Patients with a prior history of anaphylaxis.
7. Patients with chronic urticaria.
8. Patients with moderate-severe atopic dermatitis.
9. Patients with clinically relevant malformations of the upper respiratory tract.
10. Patients who have participated in another clinical trial within 3 months prior to this study.
11. Patients being treated with tricyclic antidepressants, psychotropic drugs, beta-blockers, or angiotensin-converting enzyme inhibitors (ACEIs).
12. Women who are pregnant or breast-feeding or are of child-bearing age and who do not agree to use adequate contraception if they are sexually active and who have not demonstrated that they have been surgically sterilized or have other means of not bearing children.
13. Patients who cannot attend study visits.
14. Patients who are uncooperative or refuse to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Alvarez Cuesta, MD, Principal Investigator — Hospital Universitario Ramón y Cajal; Santiago Quirce, MD, Principal Investigator — Hospital Universitario La Paz; Matilde Rodríguez, MD, Principal Investigator — Hospital Universitario Puerta de Hierro; José Manuel Zubeldia, MD, Principal Investigator — Hospital Universitario Gregorio Marañón; Carmen Panizo, MD, Principal Investigator — Hospital Ntra. Sra. del Prado; João Fonseca, MD, Principal Investigator — Instituto CUF Porto; José Luís Plácido, MD, Principal Investigator — Centro Hospitalar de S. João; José Alberto Ferreira, MD, Principal Investigator — Centro Hospitalar Gaia/Espinho; Celso Pereira, MD, Principal Investigator — Hospital da Universidade de Coimbra; Filipe Inácio, MD, Principal Investigator — Centro Hospitalar de Setúbal - Hospital de São Bernardo
Locations (10):
- Portugal (5):
  - Hospital da Universidade de Coimbra, Coimbra
  - Centro Hospitalar de S. João, Porto
  - Instituto CUF Porto, Senhora da Hora
  - Centro Hospitalar de Setúbal - Hospital de São Bernardo, Setúbal
  - Centro Hospitalar Gaia/Espinho, Vila Nova de Gaia
- Spain (5):
  - Hospital Ntra. Sra. del Prado, Talavera de la Reina, Toledo
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allergovac Depot Group 1 Active | Allergovac Depot Group 2 Active | Allergovac Depot Group 3 Active | Allergovac Depot Group 4 Active | Allergovac Depot Group 5 Active | Placebo - Group 6
Started | 27 | 25 | 24 | 24 | 25 | 26
Completed | 24 | 23 | 24 | 19 | 18 | 23
Not Completed | 3 | 2 | 0 | 5 | 7 | 3
Not completed — Protocol Violation | 2 | 2 | 0 | 3 | 1 | 1
Not completed — Change site living | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergovac Depot Group 1 Active | Allergovac Depot Group 2 Active | Allergovac Depot Group 3 Active | Allergovac Depot Group 4 Active | Allergovac Depot Group 5 Active | Placebo - Group 6 | Total
Number analyzed (Participants) | 27 | 25 | 24 | 24 | 25 | 26 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (7.7) | 31.8 (9.9) | 34.8 (9.0) | 33.5 (9.4) | 34.9 (8.3) | 35.0 (10) | 32.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 16 | 10 | 12 | 15 | 88
  Male | 9 | 8 | 8 | 14 | 13 | 11 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 9 | 7 | 8 | 8 | 54
  Not Hispanic or Latino | 15 | 15 | 15 | 17 | 17 | 18 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Variation of the Concentration of Phleum Pratense Extract Needed to Produce a Positive Nasal Provocation Test From Baseline (V0) to Final Visit (FV).
Description: Variation of the concentration of Phleum pratense extract needed to produce a positive nasal provocation test from baseline (V0) to final visit (FV). The changes will be compared among groups (including the placebo group).
Time Frame: Baseline (V0) and Final Visit (FV). The Final Visit will be conducted within 7 plus minus 2 days after the last dose is administered. The study will be carried out outside the pollination season of Phleum pratense.
Population: Intent-to-treat population (ITT): This population included all randomized patients who received at least one treatment dose and who presented baseline and post-baseline values for the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: SPT
Arm/Group | Allergovac Depot Group 1 Active | Allergovac Depot Group 2 Active | Allergovac Depot Group 3 Active | Allergovac Depot Group 4 Active | Allergovac Depot Group 5 Active | Placebo - Group 6
Number analyzed (Participants) | 25 | 25 | 24 | 23 | 23 | 23
SPT | 0.493 (2.060) | 0.275 (2.884) | 0.693 (2.142) | 0.876 (2.414) | 1.385 (2.170) | 0.839 (2.328)

2. Secondary Outcome: All Adverse Reactions and or Events Will be Recorded Both by the Patient and the Health Care Personnel Responsible for the Administration of the Subcutaneous Immunotherapy.
Description: All adverse reactions and/or events were recorded both by the patient and the health care personnel responsible for the administration of the subcutaneous immunotherapy. The incidence and intensity of adverse events was compared among the treatment groups.
Time Frame: From baseline (V0) to final visit (VF). The Final Visit will be conducted within 7 plus minus 2 days after the last dose is administered. All AE should be monitored until they are satisfactorily resolved or stabilized after the final visit of the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each participant in the research, the treatment duration was established at 17 weeks, of which 5 weeks were needed for the induction phase and the other 12 weeks were for treatment at the maintenance dose. During this period adverse event data were collected.
Description: Any unfavorable medical occurrence, including any abnormal sign (for example, abnormal physical exam), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participation in the research.
  Adverse reactions were classified as local or systemic in relation to where the reaction appeared. Local reactions appeared in the same place of administration and systemic reactions occurred far from the administration point.
Arm/Group | Allergovac Depot Group 1 Active | Allergovac Depot Group 2 Active | Allergovac Depot Group 3 Active | Allergovac Depot Group 4 Active | Allergovac Depot Group 5 Active | Placebo - Group 6
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/24 | 0/24 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/25 | 2/24 | 3/24 | 8/25 | 1/26
Other Adverse Events (participants affected / at risk) | 8/27 | 15/25 | 7/24 | 3/24 | 3/25 | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allergovac Depot Group 1 Active (N=27) | Allergovac Depot Group 2 Active (N=25) | Allergovac Depot Group 3 Active (N=24) | Allergovac Depot Group 4 Active (N=24) | Allergovac Depot Group 5 Active (N=25) | Placebo - Group 6 (N=26)
Generalized urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
cutaneous pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
generalized pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hand fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allergovac Depot Group 1 Active (N=27) | Allergovac Depot Group 2 Active (N=25) | Allergovac Depot Group 3 Active (N=24) | Allergovac Depot Group 4 Active (N=24) | Allergovac Depot Group 5 Active (N=25) | Placebo - Group 6 (N=26)
nasopharyngitis (Infections and infestations) | 6 (7) | 5 (7) | 3 (4) | 1 (1) | 1 (1) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 6 (9) | 4 (9) | 1 (1) | 1 (1) | 1 (1)
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The small simple size, the strong placebo effect and patients without a positive result with any of the tested vials at the final visit were assigned the vial 4 value for analysis purposes, meaning no real improvement could be observed in patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No